CLINICAL TRIAL: NCT00362882
Title: Randomized Phase II Trial of Sequential Versus Concurrent Docetaxel and PS-341 (NSC 681239) in Previously Treated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Docetaxel and Bortezomib in Treating Patients With Progressive or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00123; PHII-70; N01CM17101 (NIH); CDR0000491470 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Bortezomib; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients receive docetaxel IV over 60 minutes on day 1 and bortezomib IV over 3-5 seconds on days 1 and 8.
  Interventions: Drug: docetaxel; Drug: bortezomib; Other: laboratory biomarker analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: pharmacological study
- Arm 2 (Experimental): Patients receive docetaxel as in arm I and bortezomib IV over 3-5 seconds on days 2 and 8.
  Interventions: Drug: docetaxel; Drug: bortezomib; Other: laboratory biomarker analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: pharmacological study

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — correlative study
Other: immunoenzyme technique — correlative study
  Other Names: immunoenzyme techniques
Other: immunohistochemistry staining method — correlative study
  Other Names: immunohistochemistry
Other: pharmacological study — correlative study
  Other Names: pharmacological studies

SUMMARY:
This trial is studying two different schedules of docetaxel and bortezomib to compare how well they work in treating patients with progressive or recurrent non-small cell lung cancer. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving docetaxel together with bortezomib may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the efficacy and tolerability of sequential vs concurrent docetaxel and bortezomib in patients with previously treated, progressive or recurrent, advanced non-small cell lung cancer (NSCLC).

SECOND OBJECTIVES:

I. To compare time to progression in patients with previously treated NSCLC treated with these regimens.

II. To compare 1-year and overall survival of patients treated with these regimens.

III. To compare the toxicity of these regimens in these patients. IV. To determine the pharmacokinetics of docetaxel in the context of this study.

TERTIARY OBJECTIVE:

I. To determine levels of expression of molecular markers regulated by docetaxel and bortezomib and correlate with clinical response and overall survival of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG performance status (0 vs 1) and number of prior chemotherapy treatments (1 vs >1). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive docetaxel IV over 60 minutes on day 1 and bortezomib IV over 3-5 seconds on days 1 and 8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive docetaxel as in arm I and bortezomib IV over 3-5 seconds on days 2 and 8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Criteria:

* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer for which the patient is currently in complete remission, or any other cancer for which the patient has been disease-free for 5 years.
* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC).
* Progressive or recurrent NSCLC after treatment with 1 prior platinum-based chemotherapy regimen for metastatic disease. Prior neoadjuvant/adjuvant chemotherapy and/or concurrent chemoradiation for early-stage disease allowed.
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas) and recovered.
* No prior docetaxel or bortezomib
* Prior epidermal growth factor receptor inhibitor therapy allowed.
* Prior paclitaxel allowed
* At least 4 weeks since prior major surgery and recovered.
* At least 2 weeks since prior and no concurrent enzyme-inducing anticonvulsants.
* No concurrent hormonal therapy, biologic therapy, or radiotherapy to measurable lesions. Concurrent palliative radiotherapy to small-field nonindicator lesions (e.g., painful bony metastases) allowed.
* Measurable disease* with >= 1 unidimensionally objectively measurable lesion, including any of the following:
* Lung mass (measurable on chest x-ray, tomograms, or CT scan)
* Enlarged lymph nodes
* Liver metastasis (measurable as a discrete focal lesion on radionuclide or CT scan, or ultrasound)
* Metastatic abdominal mass (measurable on CT scan with >= 1 perpendicular diameter ≥ the distance between cuts)
* Measurable disease must be outside the previous radiation field or a new lesion must be present.
* Life expectancy >= 12 weeks
* Progressive disease within a previously radiated field allowed.
* [Note: *Measurable disease DOES NOT include bone metastases or non-focal liver metastases].
* No symptomatic or untreated brain metastasis requiring steroids. Asymptomatic, previously treated (surgical resection or radiotherapy) brain metastasis allowed provided they are neurologically stable and >= 4 weeks since prior steroids.
* Creatinine clearance >= 50 mL/min
* Creatinine =< 1.6 mg/dL
* Bilirubin normal
* AST =< 2 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy >= grade 2
* Absolute granulocyte count >= 1,500/mm³
* Platelet count >= 100,000/mm³
* Cutaneous nodule
* ECOG performance status 0-1
* At least 4 weeks since prior radiotherapy and recovered.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo Lara, Principal Investigator — University of California, Davis
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients receive docetaxel IV at 75 mg/m2 on day 1 and bortezomib IV at 1.6 mg/m2 seconds on days 1 and 8.
  docetaxel: Given IV
  bortezomib: Given IV
  laboratory biomarker analysis: correlative study
  immunoenzyme technique: correlative study
  immunohistochemistry staining method: correlative study
  pharmacological study: correlative study
- Arm 2: Patients receive docetaxel IV at 75 mg/m2 on day 1 and bortezomib IV at 1.6 mg/m2 seconds on days 2 and 8.
  docetaxel: Given IV
  bortezomib: Given IV
  laboratory biomarker analysis: correlative study
  immunoenzyme technique: correlative study
  immunohistochemistry staining method: correlative study
  pharmacological study: correlative study
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Median (Full Range); unit: years] | 61 [45 to 79] | 61 [32 to 82] | 61 [32 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 23 | 20 | 43
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasion | 32 | 33 | 65
  Asian | 3 | 6 | 9
  African Americian | 5 | 1 | 6
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT, MRI or X-ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 40 | 41
percentage of participants | 10 | 10

2. Secondary Outcome: Overall Survival
Description: Will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: From first day of treatment to time of death due to any cause, up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 40 | 41
Months | 13.3 [7 to 17] | 7.8 [6 to 18]

3. Secondary Outcome: Disease Control Rate
Description: Disease control rate was defined as the rate of partial response (PR) plus stable disease (SD; for at least 2 cycles).
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 40 | 41
percentage of participants | 50 | 49

4. Secondary Outcome: Progression-free Survival @ 6 Months
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Measure: Number; unit: percent of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 40 | 41
percent of participants | 30 | 17
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.17, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events reported over a period of 4 years, 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 15/40 | 21/41
Other Adverse Events (participants affected / at risk) | 40/40 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=40) | Arm 2 (N=41)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Death (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 2 (2) | 4 (4)
Fever (General disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 1 (1)
Leukopenia (Investigations) | 2 (2) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5) | 7 (7)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=40) | Arm 2 (N=41)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 29 (94) | 28 (83)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (5) | 4 (9)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (8)
Dry eye syndrome (Eye disorders) | 1 (3) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 3 (3)
Vision blurred (Eye disorders) | 2 (3) | 2 (2)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 5 (14) | 3 (5)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 12 (16)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (21) | 17 (23)
Diarrhea (Gastrointestinal disorders) | 13 (17) | 13 (15)
Dyspepsia (Gastrointestinal disorders) | 3 (9) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (4) | 5 (7)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (31) | 19 (31)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (12) | 15 (22)
Chest pain (General disorders) | 3 (3) | 3 (4)
Chills (General disorders) | 2 (3) | 2 (3)
Disease progression (General disorders) | 24 (24) | 24 (24)
Edema limbs (General disorders) | 8 (18) | 9 (12)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 30 (100) | 29 (81)
Fever (General disorders) | 4 (5) | 5 (8)
Gait abnormal (General disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 3 (4)
Pain (General disorders) | 2 (2) | 4 (6)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 1 (2) | 1 (2)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (6) | 0 (0)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (10) | 4 (5)
Alkaline phosphatase increased (Investigations) | 7 (15) | 14 (29)
Aspartate aminotransferase increased (Investigations) | 8 (24) | 7 (14)
Bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 3 (4)
Haptoglobin decreased (Investigations) | 0 (0) | 2 (2)
Hypercholesterolemia (Investigations) | 0 (0) | 1 (6)
INR increased (Investigations) | 2 (2) | 1 (2)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (2)
Leukocyte count decreased (Investigations) | 9 (17) | 13 (28)
Leukopenia (Investigations) | 5 (16) | 5 (10)
Lymphocyte count decreased (Investigations) | 15 (50) | 13 (39)
Lymphopenia (Investigations) | 7 (23) | 8 (21)
Neutrophil count decreased (Investigations) | 10 (13) | 17 (27)
Platelet count decreased (Investigations) | 10 (28) | 19 (46)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 3 (4) | 0 (0)
Weight loss (Investigations) | 1 (2) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 9 (22) | 9 (13)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 14 (39) | 16 (36)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (6) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (12) | 6 (16)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (7) | 4 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 10 (22) | 14 (22)
Serum calcium decreased (Metabolism and nutrition disorders) | 9 (14) | 3 (3)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (3) | 4 (4)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (3) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (5) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (9) | 8 (11)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (22) | 16 (32)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (16) | 5 (13)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 7 (13) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (11) | 4 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (11) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (5)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (7)
Dizziness (Nervous system disorders) | 6 (6) | 9 (11)
Headache (Nervous system disorders) | 4 (5) | 13 (17)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (41) | 11 (28)
Phrenic nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 4 (9) | 6 (6)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2) | 2 (3)
Anxiety (Psychiatric disorders) | 5 (10) | 4 (5)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 2 (9)
Insomnia (Psychiatric disorders) | 4 (9) | 10 (19)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (9)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (26) | 19 (41)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (31) | 21 (44)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (39) | 14 (41)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (5)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Flushing (Vascular disorders) | 2 (2) | 2 (3)
Hemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (3) | 2 (8)
Hypotension (Vascular disorders) | 2 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less